CLINICAL TRIAL: NCT02329262
Title: A Skills-based RCT for Physical Activity Using Peer Mentors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Laureen Smith, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014B0094
Record Dates: First submitted 2014-12-17; First posted 2014-12-31 (Estimated); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Health Behavior; Obesity; Motor Activity
Keywords: exercise; mentors; health education; obesity
MeSH Terms: conditions — Health Behavior; Obesity; Motor Activity; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mentoring to be Active (Experimental): Trained teen mentors will deliver the physical activity curriculum to high school students in a school setting. Physical activity will be measured with accelerometers.
  Interventions: Behavioral: Mentoring to be Active with Accelerometers
- Planning to be Active (Active Comparator): High school teachers will deliver the physical activity curriculum (usual care) to high school students enrolled in health education courses. Physical activity will be measured with accelerometers.
  Interventions: Behavioral: Planning to be Active with Accelerometers
- Peer Mentors (No Intervention): 11 and 12 grade-level trained mentors who lead the Mentoring to be Active (MBA) experimental group as peer mentors.
- High School Teachers (No Intervention): High School teachers who taught the usual care healh classes for the Planning to be Active (PBA) active comparator group.

INTERVENTIONS:
Behavioral: Mentoring to be Active with Accelerometers — Trained high school mentors will deliver a 10 session curriculum targeting physical activity to younger teens.
  Other Names: peer mentoring
  Arms: Mentoring to be Active
Behavioral: Planning to be Active with Accelerometers — Health education teachers will deliver the 10 session curriculum targeting physical activity to high school students enrolled in health courses.
  Other Names: Teacher PBA
  Arms: Planning to be Active

SUMMARY:
This approach will train peer mentors to deliver a culturally appropriate intervention and provide social support that is critical for facilitating and sustaining health behavior change. The objective is to compare the efficacy of an innovative healthy lifestyle skills mentoring program (Mentored Planning to be Active [MBA]) to a teacher led program (PBA) for increasing physical activity in Appalachian high school teens. MBA emphasizes the social determinants of health by using a social networking approach that trains peer mentors to support targeted teens

DETAILED DESCRIPTION:
The goal of this study is to positively impact the physical activity patterns to improve health outcomes including the high rates of obesity in Appalachian teens. The approach will train peer mentors to deliver the culturally appropriate intervention and provide social support that is critical for facilitating and sustaining health behavior change. The primary objective is to compare the efficacy of an innovative healthy lifestyle skills mentoring program (Mentored Planning to be Active [MBA]) to a teacher led program (PBA) for increasing physical activity in Appalachian high school teens. MBA emphasizes the social determinants of health by using a social networking approach that trains peer mentors to support targeted teens. Refined over the course of 3 studies,2-4 PBA is a ten-lesson unit delivered over 10 weeks and designed to teach self-regulation of physical activity among teens. Expanding PBA to mentors via MBA has the potential to promote and sustain adoption of daily regular physical activity through self-regulation of physical activity in discretionary time. With MBA delivery, physical activity is tailored to personal interests, talents, and neighborhood environment. MBA empowers students to plan and evaluate their own personal activity plan. It is predicted that by serving as role models, peer mentors will improve their own lifestyle behaviors, providing a double-edged intervention. It is also predicted that providing intense and structured social support to teens via peer mentors will result in better health outcomes compared to teacher-based support alone (usual care). The plan is to conduct a group randomized controlled trial to evaluate the effects of a culturally and theoretically based behavioral intervention delivered by peer mentors (MBA) on adolescent healthy behaviors (daily physical activity, regular exercise, and sedentary behaviors) and physical health outcomes (BMI, body fat) compared to PBA delivered in a classroom setting by a teacher.

ELIGIBILITY:
Inclusion Criteria:

* 9th or 10th grade students as participants
* 11th or 12th grade students as mentors
* Classroom teachers who instruct health education or physical education to 9th and 10th grade students.
* Not expected to move from school prior to conclusion of study
* Speaks English

Exclusion Criteria:

* Peer mentors with a BMI (for age and gender) above the 85th percentile or below the 5th percentile at the start of the study

Ages: 14 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 571 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laureen H Smith, PhD, Principal Investigator — OSU College of Nursing; Rick L Petosa, PhD, Principal Investigator — Ohio State University
Locations (20):
- United States (20):
  - River Valley High School, Bidwell, Ohio
  - Chillicothe High School, Chillicothe, Ohio
  - Huntington Local High School, Chillicothe, Ohio
  - Unioto High School, Chillicothe, Ohio
  - Zane Trace High School, Chillicothe, Ohio
  - Dawson-Bryant High School, Coal Grove, Ohio
  - Green High School, Franklin Furnace, Ohio
  - Ironton High School, Ironton, Ohio
  - Jackson High School, Jackson, Ohio
  - Western High School, Latham, Ohio
  - New Boston High School, New Boston, Ohio
  - Oak Hill High School, Oak Hill, Ohio
  - Piketon High School, Piketon, Ohio
  - Clay Local High School, Portsmouth, Ohio
  - West Portsmouth High School, Portsmouth, Ohio
  - Southern Local High School, Racine, Ohio
  - South Point High School, South Point, Ohio
  - Federal Hocking High School, Stewart, Ohio
  - Berne Union High School, Sugar Grove, Ohio
  - Waverly High School, Waverly, Ohio

REFERENCES:
- [Background] Smith LH, Petosa RL. A Structured Peer-Mentoring Method for Physical Activity Behavior Change Among Adolescents. J Sch Nurs. 2016 Oct;32(5):315-23. doi: 10.1177/1059840516644955. Epub 2016 May 4. PMID 27257081
- [Background] Smith LH, Petosa RL. Effective Practices to Improve Recruitment, Retention, and Partnerships in School-Based Studies. J Pediatr Health Care. 2016 Sep-Oct;30(5):495-8. doi: 10.1016/j.pedhc.2016.05.004. Epub 2016 Jun 16. No abstract available. PMID 27321677
- [Derived] Smith LH, Petosa RL, Shoben A. Peer mentor versus teacher delivery of a physical activity program on the effects of BMI and daily activity: protocol of a school-based group randomized controlled trial in Appalachia. BMC Public Health. 2018 May 16;18(1):633. doi: 10.1186/s12889-018-5537-z. PMID 29769106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: students attending the same school are expected to socialize together; thus, a Group-Randomized Control Trial (G-RCT) is necessary to avoid the risk of cross-contamination.There were 20 high schools recruited in 3 waves, with 4 in Wave 1, 8 in Wave 2, and 8 in Wave 3, for a total of schools. For each wave of schools, half of the schools were randomly assigned to each condition-intervention [MBA] and comparison [PBA]-for a total of 10 schools in each of the two conditions by study's end.
Units Other Than Participants: schools
Groups:
- Mentoring to be Active (MBA): Trained teen mentors delivered the physical activity curriculum to younger high school students in a school setting. Physical activity was measured with accelerometers. Data not collected from peer mentors.
  Mentoring to be Active with Accelerometers: Trained high school mentors delivered a 10-session curriculum targeting physical activity to younger teens.
- Planning to be Active (Usual Care): High school teachers delivered the physical activity curriculum (usual care) to high school students enrolled in health education courses. Physical activity was measured with accelerometers.
  Planning to be Active with Accelerometers: Health education teachers will delivered the 10-session curriculum targeting physical activity to high school students enrolled in health courses.
Period: Overall Study
Arm/Group | Mentoring to be Active (MBA) | Planning to be Active (Usual Care)
Started (Total participants) | 318; 10 schools | 253; 10 schools (Data not collected from classroom teachers.)
Student Participants | 252; 10 schools | 248; 10 schools
Peer Mentors (11th and 12th grade level trained mentors who lead the Mentoring to be Active (MBA) as intervention specialists.) | 66; 0 schools | 0; 0 schools
Teachers (High School teachers who taught the usual care health classes. Data not collected from classroom teachers.) | 0; 0 schools | 5; 0 schools
Completed | 318; 10 schools | 253; 10 schools
Not Completed | 0; 0 schools | 0; 0 schools

BASELINE CHARACTERISTICS:
Population: The participant population is consistent with the overall population demographics of the counties that the schools are located in.
Groups:
- Mentoring to be Active: Trained teen mentors will deliver the 10- session physical activity curriculum to high school students in a school setting. Physical activity will be measured with accelerometers.
- Planning to be Active: High school teachers will deliver the 10- session physical activity curriculum (usual care) to high school students enrolled in health education courses. Physical activity will be measured with accelerometers.
- Peer Mentors: 11th and 12th grade level trained mentors who lead the Mentoring to be Active (MBA) as intervention specialists
- High School Teachers: High School teachers who taught the usual care health classes.
- Total: Total of all reporting groups
Arm/Group | Mentoring to be Active | Planning to be Active | Peer Mentors | High School Teachers | Total
Number analyzed (Participants) | 252 | 248 | 66 | 5 | 571
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 252 | 248 | 66 | 0 | 566
  Between 18 and 65 years | 0 | 0 | 0 | 5 | 5
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 14.84 [13 to 16] | 15.25 [13 to 16] | 16.49 [15 to 17] | 38.38 [32 to 44] | 14.97 [13 to 16]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 122 | 122 | 27 | 3 | 274
  Female | 130 | 126 | 39 | 2 | 297
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 3 | 0 | 5
  Not Hispanic or Latino | 251 | 247 | 63 | 4 | 565
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15 | 11 | 0 | 0 | 26
  Asian | 5 | 1 | 2 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 13 | 4 | 1 | 28
  White | 222 | 219 | 56 | 3 | 500
  More than one race | 0 | 4 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 252 | 248 | 66 | 5 | 627
Grade level at beginning of study [Count of Participants; unit: Participants]
  9th grade | 252 | 248 | 0 | 0 | 500
  10th grade | 0 | 0 | 2 | 0 | 2
  11th-12th gradee | 0 | 0 | 64 | 0 | 64
  N/A | 0 | 0 | 0 | 5 | 5
Average Number of Household Members [Mean (Standard Deviation); unit: number of household members] — Number of persons living in the primary residence with the participant. Number indicates additional persone living with the participant.
  number of household members | 4.3 (3.9) | 4.6 (3.5) | 4.5 (3.2) | 5.2 (2.8) | 4.4 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index From T1 to T3
Description: Body mass index is caculated as weight in kilograms divided by the square of height in meters.
  The measure is the change in BMI from baseline to 9 months post-baseline.
Time Frame: T1 (Baseline) to T3 (9 months-post baseline)
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Mentoring to be Active | Planning to be Active
Number analyzed (Participants) | 252 | 248
kg/m2 | -.9257 (1.76) | -.6503 (2.09)

2. Primary Outcome: Change in Total Body Weight From T1 to T3
Description: Change in total body weight from baseline to 9 months post-baseline.
Time Frame: T1 (baseline) to T3 (9-month post baseline)
Measure: Mean (Standard Deviation); unit: pounds
Groups:
- Planning to be Active: Eight high school teachers delivered the physical activity curriculum (usual care) to 248 high school students enrolled in health education courses. Physical activity was measured with accelerometers. Baseline data not collected from teachers.
- Mentoring to be Active: Peer mentors delivered the 10-session curriculum to 252 students.
Arm/Group | Planning to be Active | Mentoring to be Active
Number analyzed (Participants) | 248 | 252
pounds | -4.96 (11.38) | 8.72 (10.94)

3. Primary Outcome: Change in Pounds of Body Fat From T1 to T3
Description: Body fat in pounds measured by Tanita Body Composition Analyzer.
  This equipment provides estimated values for each measured value of body fat percentage, fat mass, fat free mass, muscle mass and bone mass by the DXA method, estimated value for the total body water measured value by the dilution method and estimated value for the visceral fat rating by MRI method using the Bioelectrical Impedance Analysis (BIA method). The Tanita Body Composition Analyzer measures body composition using a constant current source with a high frequency current (6.25kHz, 50kHz, 90μA). The 4 electrodes are positioned so that electric current is supplied from the electrodes on the tips of the toes of both feet, and voltage is measured on the heel of both feet. Body weight measured with shoes and socks removed. Calculated to the nearest 0.2 pounds.
Time Frame: T1 ( Baseline) to T3 (9-months post baseline)
Measure: Mean (Standard Deviation); unit: pounds
Groups:
- Planning to be Active: Eight high school teachers delivered the physical activity curriculum (usual care) to 248 high school students enrolled in health education courses. Physical activity was measured with accelerometers. Baseline data not collected from teachers.
  Planning to be Active with Accelerometers: Health education teachers will delivered the 10-session curriculum targeting physical activity to high school students enrolled in health courses.
Arm/Group | Planning to be Active | Mentoring to be Active
Number analyzed (Participants) | 248 | 252
pounds | -3.05 (11.46) | -3.13 (12.44)

4. Secondary Outcome: Moderate Physical Activity (Daily)
Description: Percentage of participants engaging in daily moderate physical activity. Measured by accelerometers; subjects to wear devices for 7 days at each data collection time point
Time Frame: 9 months
Measure: Number; unit: percentage of participants
Arm/Group | Mentoring to be Active | Planning to be Active
Number analyzed (Participants) | 252 | 248
percentage of participants | 4.9 | 4.9

5. Secondary Outcome: Outcome Expectancies Scale
Description: 21 item, 6 -point Likert Summative Scale focusing on psychological determinants of physical activity. Higher values indicate higher (more positive) outcome expectancies. Range of scores are from 21-126 with a score of 63 or higher indicating more positive expectancy from engaging in physical activity.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mentoring to be Active | Planning to be Active
Number analyzed (Participants) | 177 | 158
score on a scale | 81.47 (13.6) | 81.8 (13.4)

6. Secondary Outcome: Exercise Self-Efficacy Scale
Description: 14 item scale that asks participants to rank their own confidence in performing an exercise behavior from 0% confidence to 100 % confidence. Higher percentages indicate higher levels of self-efficacy to engage in physical activity. Each item may range from 0% to 100%. An item score of 51% indicates "positive" confidence. Eight or more items with at least 51% for each indicates overall" positive self-efficacy" to engage in exercise. The total scale may range from 0 (no confidence)-1400 (100% confidence on each item). A score of 408 or higher (at least 51% on a minimum of 8/14 items) indicates "positive" self-efficacy to engage in exercise.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mentoring to be Active | Planning to be Active
Number analyzed (Participants) | 183 | 172
score on a scale | 783 (304) | 830 (315)

7. Secondary Outcome: Outcome Expectations Scale
Description: 40 item, 6-point Likert type scale that asks participants to rank their expectations of what physical activity will do their own health outcomes. Scores range from 40-240. Scores of 101 or above indicate more positive expectation of what physical activity can do to health outcomes (more positive health outcomes expected)
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mentoring to be Active | Planning to be Active
Number analyzed (Participants) | 175 | 167
score on a scale | 68.5 (12.9) | 70.3 (13.8)

8. Secondary Outcome: Social Support From Family and Friends to Exercise
Description: 12 item, 5 point Likert measure asking participants to rate each question twice: Once for family members and once for friends. Questions ask about the perceived social support to engage in physical activity within the past 3 months. Higher values indicate more social support to engage in physical activity. Values range from 12-60 for the Family Social Support and 12-60 for Friends Social Support. A total social support score is created by summing the scores for family and friends combined. A total score of 25 or above for indicates higher or more positive social support.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mentoring to be Active | Planning to be Active
Number analyzed (Participants) | 178 | 163
score on a scale | 29.4 (13.3) | 33.2 (13.9)

9. Secondary Outcome: Vigorous Physical Activity
Description: Percentage of participants engaging in vigorous physical activity during the data collection period measured by accelerometers.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Groups:
- Mentoring to be Active: Trained teen mentors (n = 129) delivered the physical activity curriculum to 252 high school students in a school setting. Physical activity was measured with accelerometers. Data not collected from peer mentors.
Arm/Group | Mentoring to be Active | Planning to be Active
Number analyzed (Participants) | 252 | 248
Participants | 176 | 198

10. Other Pre Specified Outcome: Sessions Attended
Description: Average number of sessions attended by participants
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Mentoring to be Active | Planning to be Active
Number analyzed (Participants) | 251 | 78
sessions | 6.98 (3.2) | 9.6 (1.1)

11. Post Hoc Outcome: Ease of Use
Description: Participants will be asked to describe the ease of using the intervention curriculum and comparison program. General satisfaction with the program will be assessed.
Time Frame: 3 months
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: Adverse event data collected during the study timeframe, from baseline through the 9-month post-baseline follow-up period.
Description: This study was minimal risk; participants engaged in activities that occur in every day life.
Arm/Group | Mentoring to be Active | Planning to be Active | Peer Mentors | High School Teachers
All-Cause Mortality (participants affected / at risk) | 0/252 | 0/248 | 0/66 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/252 | 0/248 | 0/66 | 0/5
Other Adverse Events (participants affected / at risk) | 0/252 | 0/248 | 0/66 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT02329262/Prot_SAP_000.pdf